CLINICAL TRIAL: NCT05644912
Title: Exploratory Investigation on a Novel Catheter
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wellspect HealthCare (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: NAV-0010
Record Dates: First submitted 2022-11-18; First posted 2022-12-09 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2023-04

CONDITIONS: Bowel Dysfunction
MeSH Terms: conditions — Intestinal Diseases

STUDY DESIGN:
Intervention Model Description: Proof of concept investigation with subjects experienced in using transanal irrigation with a balloon catheter.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All subjects (Experimental): Transanal irrigation (TAI) with new catheter
  Interventions: Device: Transanal irrigation (TAI)

INTERVENTIONS:
Device: Transanal irrigation (TAI) — Transanal irrigation (TAI) with new catheter on subjects experienced in using TAI with balloon catheter.

SUMMARY:
An exploratory, pre-market, open, prospective, interventional, clinical investigation at a limited number of centers for proof of concept of a new catheter.

In this proof of concept investigation, subjects experienced in using transanal irrigation (TAI) with a balloon catheter will be using study catheters at two occasions to primarily study if the catheter will stay in place during the water instillation when performing TAI.

Each subject will be followed during approximately one week, depending on the usual time between their TAI.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of informed consent.
2. Female and male aged 18-80 years.
3. Patients successfully treated by TAI with Navina Smart system for at least 3 months and/or stable in therapy.
4. Patients considered suitable to participate by investigator.
5. Able to read, write and understand information given to them regarding the study.

Exclusion Criteria:

1. Involvement in the planning and conduct of the clinical investigation (applies to both Wellspect HealthCare staff and staff at the study site).
2. Previous enrolment in the present clinical investigation.
3. Simultaneous participation in another clinical investigation, or participation in a clinical investigation during the last month, that may interfere with the present clinical investigation.
4. Severe non-compliance to Clinical Investigation Plan as judged by the investigator and/or Wellspect HealthCare.
5. Significant cardiovascular and/or other significant co-morbidities which could be negatively affected by the use of the investigational product.
6. Known anal or colorectal stenosis.
7. Active inflammatory bowel disease.
8. Acute diverticulitis.
9. Colorectal cancer.
10. Ischemic colitis.
11. Any anal or colorectal surgery within the previous 3 months.
12. Anal, rectal and/or colonic endoscopic polypectomy within the previous 4 weeks.
13. Any condition, as judged by the investigator, which might make follow-up or investigations inappropriate.
14. Any patient that according to the Declaration of Helsinki is unsuitable for enrolment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2022-11-18 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2023-12-15 (Actual)

PRIMARY OUTCOMES:
Catheter stay in place | 1 week
  Does the catheter stay in place during water instillation? Yes/No

SECONDARY OUTCOMES:
Bowel emptying performance | 1 week
  Evaluation of bowel emptying performance: Subject's perception of emptying of bowel similar to regular use of TAI.
  Descriptive analysis of data from questionnaires at Visit 2 and 3 collected from subject's previous experience from using balloon catheter comparing it with experience of using two different sizes of study catheters during study.
  Question asked: "What is the subject's perception of emptying of bowel with the study catheter compared to their regular use with a balloon catheter?" Potential response: much worse, worse, same, better, much better
Leakage | 1 week
  Evaluation of leakage during water instillation: Subject's perception of leakage similar to regular use of TAI.
  Descriptive analysis of data from questionnaires at Visit 2 and 3 collected from subject's previous experience from using balloon catheter comparing it with experience of using two different sizes of study catheters during study.
  Question asked: "What is the subject's perception of leakage with the study catheter compared to their regular use with a balloon catheter?" Potential response: much worse, worse, same, better, much better

OTHER OUTCOMES:
Safety: Adverse Events and Device Deficiencies | 1 week
  To evaluate the safety of catheter by assessment of incidence and severity of Adverse Events (AEs, SAEs, ADEs, SADEs, USADEs) and Device Deficiencies occurring during the study period.

CONTACTS AND LOCATIONS:
Overall Officials: Ingrid Han-Geurts, MD, Principal Investigator — Proctos Kliniek
Locations (1):
- Proctos Kliniek, Bilthoven, MB Bilthoven, Netherlands

IPD SHARING:
Plan to Share IPD: No
IPD available will not be available to other researchers.